CLINICAL TRIAL: NCT03889951
Title: Detection of IKZF1 Deletion Mutation in Patients With Acute Lymphoblastic Leukemia and Its Impact in Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin Tarek Elgammal, principal investigator, Assiut University
Other Study IDs: ikzf1 in all
Record Dates: First submitted 2019-02-28; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: ALL, Childhood
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1: group of ALL patients with IKZF1 deletion mutation.
- group 2: group of ALL patients with no detected mutation

SUMMARY:
1. To detect IKZF-1 deletion mutations in patients with ALL.
2. To study the impact of IKZF-1 deletion mutation on therapy of ALL.
3. To study the correlation between IKZF-1 deletion mutations and BCR-ABL.

DETAILED DESCRIPTION:
Acute lymphoblastic leukemia (ALL) a malignant transformation and proliferation of lymphoid progenitor cells in the bone marrow, blood and extramedullary sites. While 80% of ALL occurs in children, it represents a devastating disease when it occurs in adults . predisposing factors include exposure to ionizing radiation, pesticides, certain solvents or viruses such as Epstein-Barr Virus and Human Immunodeficiency Virus. However, in the majority of cases, it appears as a de novo malignancy in previously healthy individuals. Chromosomal aberrations are the hallmark of ALL, but are not sufficient to generate leukemia. Characteristic translocations include t(12;21) [ETV6-RUNX1], t(1;19) [TCF3-PBX1], t(9;22) [BCR-ABL1] . More recently, a variant with a similar gene expression profile to (Philadelphia) Ph-positive ALL but without the BCR-ABL1 rearrangement has been identified. In more than 80% of cases of this so-called Ph-like ALL, the variant possesses deletions in key transcription factors involved in B-cell development including IKAROS family zinc finger 1 (IKZF1) . IKZF1 codes Ikaros, which is a member of a family of zinc- finger nuclear proteins that is required for the earliest stages of lymphoid lineage commitment and acts as tumor suppressor. Most IKZF1 mutations (94%) are deletion mutations, and there are rare point mutations resulting in loss of function of Ikaros .

There are two major deletions occur in the IKZF1 gene:

* The first one was characterized by loss of exons 4 to 7 ( 4-7) with breakpoints occurring in introns 3 and 7 on chromosome 7p12.
* The second deletion involved exons 2 to 7 ( 2-7) with a variable pattern of breakpoints in intron 1 and intron 7 in the same region as those of the 4-7 deletion.

IKZF1 mutations in cases of B-ALL are associated with poor prognosis and high risk of relapse. IKZF1 mutations are found in approximately 15% to 20% of pediatric B-ALL cases and in >75% of pediatric BCR-ABL positive ALL cases. The incidences of IKZF1 mutations in adults are approximately 50% in B-ALL cases and approximately 65% in BCR-ABL positive ALL cases .

The presence of either IKZF1 mutation or BCR- ABL has been reported to be an independent risk factor of poor prognosis for patients with B-ALL .

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute lymphoblastic leukemia.

Exclusion Criteria:

* patients with any other hematological malignancies.
* patients receiving chemotherapy.

Ages: 1 Year to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients newly diagnosed with acute lymphoblastic leukemia age ranged from 1 year to 70 years.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
detection of IKZF-1 deletion mutations in patients with ALL. | baseline
  detection of IKZF1 deletion mutation by fluorescent inset hybridization and by PCR.
Detection of BCR-ABL translocation. | baseline
  by PCR